CLINICAL TRIAL: NCT03200288
Title: A Phase 3,Randomized,Double-blind,Placebo-controlled Study to Evaluate the Clinical Performance and Safety of an Intra-articular Solution of High and Low Molecular Weight Hyaluronic Acid (HL-01) in the Treatment of Pain in Symptomatic Knee Osteoarthritis
Brief Title: A Study to Evaluate the Clinical Performance and Safety of an Intra-articular Hyaluronic Acid in Knee Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IBSA Institut Biochimique SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16EU-Hai13
Record Dates: First submitted 2017-06-21; First posted 2017-06-27 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2019-02

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: During the course of the study only the physicians who will perform the intra-articular injection (injectors) will be unblinded. All the other physicians (assessors) and study participants will be blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HL-01 (Experimental): Single 2 ml intra-articular injection of HL-01 (solution of high and low molecular weight hyaluronic acid (HA))
  Interventions: Device: HL-01: high and low molecular weight hyaluronic acid
- Placebo (Placebo Comparator): Single 2 ml intra-articular injection of Placebo (physiological solution)
  Interventions: Device: Placebo

INTERVENTIONS:
Device: HL-01: high and low molecular weight hyaluronic acid — 2 ml intra-articular single injection
  Other Names: Sinovial HL®
  Arms: HL-01
Device: Placebo — 2 ml intra-articular single injection
  Arms: Placebo

SUMMARY:
This is a study to evaluate the Clinical Performance and Safety of a single intra-articular (i.a.) injection of hyaluronic acid product (as HL-01) in the treatment of pain due to osteoarthritis (OA) of the knee.

ELIGIBILITY:
Inclusion Criteria:

* Female and male subjects ≥40 to 80 years of age.
* Subjects with primary knee OA of the medial or lateral femoro-tibial compartment, documented according to ACR criteria with symptoms, at screening, from at least 3 months.
* Subjects with Kellgren & Lawrence (K-L) radiological grade 2-3.
* Subjects with at least one antero-posterior view X-Ray image of the target knee taken within 12 months prior to the screening.
* Subjects with OA pain intensity meeting the criteria below:

If unilateral knee OA: Subjects demonstrating at screening pain intensity in the target knee measured by Visual Analogue Scale (VAS) ≥40 mm VAS, and ≤ 20 mm in the contralateral knee and confirmed at randomization after wash-out from analgesics/NSAIDs.

If bilateral knee OA: definition of the most symptomatic joint at screening based on subject's evaluation and Investigator's clinical judgment with subjects demonstrating pain intensity in the target knee measured by Visual Analogue Scale (VAS) ≥40 mm VAS, and ≤ 20mm in the contralateral knee and confirmed at randomization after wash-out from analgesics/NSAIDs.

* Subjects are able to understand and are willing and able to comply with study procedures including usage of acetaminophen as the only analgesic.
* Subjects are able to provide informed consent.
* Any female subject of childbearing potential must agree to use adequate methods of contraception throughout the course of the study.

Exclusion Criteria:

* Subjects with secondary (post-traumatic) knee OA of the target and non-target joints.
* Subjects with K-L radiological grade 4 knee OA.
* Subjects with a history of knee joint replacement/arthroplasty of the target knee.
* Subjects with a history of arthroscopy, osteotomy, or surgery of the target knee in the past 12 months.
* Subjects with any significant injury to the target knee in the last 6 months (as per Investigator judgment).
* Subjects with Body Mass Index (BMI) ≥32 kg/m2.
* Subjects with any musculoskeletal condition affecting the target knee that would impair proper assessment of the Investigational Medicinal Device (IMD) performance in the target knee as assessed by the Investigator and such as:

  1. severe varus/valgus deformity (>15°)
  2. predominantly patello-femoral pain/syndrome.
* Subjects with a history of symptomatic hip OA or other health condition i.e. associated with pain and interfering with adequate study endpoints evaluation.
* Subjects with a known history or present evidence of conditions which may affect the target knee assessments, like rheumatic disease and inflammatory, infective or metabolic joint diseases; recurrent clinical chondrocalcinosis; crystal arthropathies; osteo-articular pathologies differing from arthrosis; articular fracture; ochronosis; acromegaly; haemochromatosis; Wilson's disease; primary osteochondromatosis; heritable disorders; collagen gene mutations.
* Subjects with venous or lymphatic stasis in the relevant limb.
* Subjects with a history of the following treatments for knee OA:

  a) I. a. knee corticosteroids: i. target knee - in the past 3 months ii. non-target knee/other joints - in the past 4 weeks b) Systemic (both oral and parenteral) and topical corticosteroids at the target knee in the past 3 months.

  c) Topical anti-inflammatories and analgesics applied at the target knee in the past 48 hrs.

  d) Viscosupplementation with hyaluronic acid or joint-lavage in the target knee in the past year.

  e) Physical therapy started in the last 3 months in the target knee. f) Symptomatic Slow-Acting Drugs for OA (SYSADOA) such as glucosamine, chondroitin sulfate, diacerhein, or other medications like avocado/soya extracts, etc. in the past 3 months.

  g) Chronic or recurrent use of narcotic analgesics. h) Use of analgesic (other than acetaminophen) and NSAIDs for a time of 5-half-lives before the screening.
* Subjects with a history of chronic or recurrent use of NSAIDs/analgesics/narcotics because of diseases different from OA of the target knee.
* Subjects treated with drugs having an influence on pain: hypnotics, muscle relaxants, anxiolytics if the intake has started less than 8 days before the screening.
* Subjects who currently use heparin or anti-vitamin K (e. g. crystalline warfarin) anticoagulant therapy.
* Subjects with the presence of infection, skin diseases, other disease or trauma in the area of the injection site or joint.
* Subjects with a known history or suspected allergy or hypersensitivity to hyaluronic acid or to hyaluronate preparations.
* Subjects with a known history or suspected allergy or hypersensitivity to acetaminophen.
* Subjects with any major surgery scheduled in the next 6 months.
* Subjects who have participated in a clinical study / investigation in the last 3 months.
* Pregnant or lactating women and women of childbearing potential not willing to use adequate contraception.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 692 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2018-06-27 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Change in VAS (Visual Analogue Scale) pain score | Baseline-week 24
  The primary efficacy variable will be the change from baseline of the VAS pain score calculated as a VAS measure ranging from 0 to 100 mm. A four- step analysis will be followed in order to assess superiority of HL-01 versus Placebo after 6, 12, 18 and 24 weeks.

SECONDARY OUTCOMES:
Change in Lequesne's Algofunctional Index | Baseline-Week 24
  Change from baseline in Lequesne's Algofunctional Index at 6, 12, 18 and 24 weeks.
Change in global status assessed by subject (EQ-5D-5L EuroQol Group Health questionnaire) | Baseline-Week 24
  Change from baseline in global status assessed by subject at 6, 12, 18 and 24 weeks (EQ-5D-5L)
Change in global status assessed by physician | Baseline -Week 24
  Change from baseline in global status assessed by physician at 6, 12, 18 and 24 weeks (5-point verbal Likert scale), dichotomised to 'Improvement' and 'No change/Worsening'
Overall response rate according to OMERACT (Outcome Measures in Rheumatology)-OARSI (Osteoarthritis Research Society International) criteria | Week 6-Week 24
  Overall response rate according to OMERACT-OARSI criteria at 6, 12, 18 and 24 weeks (this is a statistical analysis)
Rescue medication usage | Week 6-Week 24
  Rescue medication usage assessed at 6, 12, 18 and 24 weeks.

OTHER OUTCOMES:
Adverse Events | Screening -Week 24
  Incidence and frequency of AEs (adverse events)
Level of treatment satisfaction | Baseline-Week 6
  Level of treatment satisfaction - assessed by subject at baseline (within 15 minutes after the i. a. injection), in 24 hours (+/- 1 hour) after the injection, at week 1 and week 6

CONTACTS AND LOCATIONS:
Locations (31):
- CHU Centre Ville (Brull) - Bone Metabolism Unit, Liège, Belgium
- Germany (4):
  - Rheumazentrum Prof. Dr. med. Gunther Neeck, Bad Doberan
  - Klinische Forschung Berlin-Mitte GmbH, Berlin
  - DGS Schmerzzentrum Eichstätt, Eichstätt
  - AmBeNet GmbHDas Ambulante BehandlungsNetz, Leipzig
- Hungary (6):
  - Revita Rendelő, Budapest
  - Semmelweis Egyetem - Ortopediai Klinika, Budapest
  - Szent Margit Rendelőintézet, Budapest
  - DEEK University, Debrecen
  - MEDIDEA Egeszsegugyi es Szolgaltato Beteti Tarsasag, Kiskunfélegyháza
  - Swan Med SMO, Létavértes
- Italy (3):
  - Istituto Ortopedico Gaetano Pini, Milan
  - Fisiatria Policlinico di Napoli, Napoli
  - Ospedale San Pietro - FATEBENEFRATELLI, Roma
- Poland (17):
  - NZOZ VITAMED Gałaj i Cichomski Sp. j., Bydgoszcz
  - ETG Chełm, Chełm
  - Centrum Medyczne Lukamed, Chojnice
  - Centrum Kliniczno-Badawcze, Elblag
  - Gdańskie Centrum Zdrowia, Gdansk
  - ETG Łódź, Lodz
  - Klinika Zdrowej Kości, Lodz
  - ETG Lublin, Lublin
  - SOLB - Zbigniew Zegota, Ostróda
  - ETG Siedlce, Siedlce
  - RCMed, Sochaczew
  - Lubelskie Centrum Diagnostyczne, Świdnik
  - ETG Warszawa, Warsaw
  - Europejskie Centrum Leczenia Chorób Cywilizacyjnych, Warsaw
  - NZOZ Wilmed, Warsaw
  - Wasilczyk Medical Clinic Indywidualna Praktyka Lekarska Cezary Wasilczyk, Warsaw
  - ETG Zamość, Zamość

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Migliore A, Blicharski T, Plebanski R, Zegota Z, Gyula G, Rannou F, Reginster JY. Knee Osteoarthritis Pain Management with an Innovative High and Low Molecular Weight Hyaluronic Acid Formulation (HA-HL): A Randomized Clinical Trial. Rheumatol Ther. 2021 Dec;8(4):1617-1636. doi: 10.1007/s40744-021-00363-3. Epub 2021 Aug 30. PMID 34462887
- [Derived] Bruyere O, Dardenne N, Donneau AF, Reginster JY. Responder Profile to Pharmaceutical-Grade Chondroitin Sulfate: An Analysis of the CONCEPT Trial. Adv Ther. 2020 Nov;37(11):4641-4648. doi: 10.1007/s12325-020-01484-x. Epub 2020 Sep 21. PMID 32954487